CLINICAL TRIAL: NCT00907244
Title: CHP-901:Arterial Spin Labeling Perfusion MR Imaging in Pediatric Brain Tumors
Brief Title: Arterial Spin Labeling Perfusion Magnetic Resonance (MR) Imaging in Pediatric Brain Tumors
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Other Study IDs: CHP 901 ASL; 2008-4-5917 (Other: Children's Hospital of Philadelphia IRB)
Record Dates: First submitted 2009-05-20; First posted 2009-05-22 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-01

CONDITIONS: Brain Tumors
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to get information regarding the usefulness and accuracy of this new magnetic resonance imaging (MRI) technique - termed arterial spin labeling (ASL) - in the diagnosis of pediatric brain tumors.

DETAILED DESCRIPTION:
The purpose of this study is to get information regarding the usefulness and accuracy of this new MRI technique - termed arterial spin labeling (ASL) - in the diagnosis of pediatric brain tumors. This technique can non-invasively measure the blood flow to the brain during MRI examination. Because aggressive brain tumors require new blood vessels and a high level of blood supply to support its growth, we believe the tumor blood flow measured using ASL is a reliable indicator of tumor grade. This information may be useful for doctors to make treatment decisions and to monitor patients' response to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-18 years
* Primary brain tumor (newly diagnosed or recurrent) with measurable disease (at least 1cm2)

Exclusion Criteria:

* Patients with cardiac pacemaker or ferrous metal foreign bodies
* Patients with medical problems contradictive to receiving MRI scans.
* Patients requiring general anesthesia or sedation for their MRI scan.
* Patients with a history of cerebrovascular disorders (stroke, moya moya) that may alter cerebral perfusion.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients between 0-18 years who are diagnosed with primary brain tumor, undergoing MRI for clinical purpose are eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2008-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fisher, M.D., Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States